CLINICAL TRIAL: NCT02186431
Title: Contact Lenses and Infiltrative Keratitis
Acronym: CLIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York College of Optometry (Other)
Responsible Party: Principal Investigator, Kathryn Richdale, Assistant Professor, State University of New York College of Optometry
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CLIK_601933
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Keratitis
Keywords: Contact lenses
MeSH Terms: conditions — Keratitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- history of corneal infiltrative events (Experimental): To quantify and compare baseline tear proteins and ocular response in contact lens wearers with a history of corneal infiltrative events
  Interventions: Device: senofilcon A
- without a history of corneal infiltrative events (Active Comparator): To quantify and compare baseline tear proteins and ocular response in contact lens wearers without a history of corneal infiltrative events.
  Interventions: Device: senofilcon A

INTERVENTIONS:
Device: senofilcon A
  Other Names: Acuvue Oasys

SUMMARY:
To quantify and compare baseline tear proteins and ocular response in contact lens wearers with a history of corneal infiltrative events, to those without a history of complications. This will be accomplished via measurement of select anti-inflammatory tear proteins before, during and after contact lens wear.

ELIGIBILITY:
Inclusion Criteria:

* Soft contact lens wearers
* Healthy (control), or with history of infiltrative keratitis (case)
* Has a wearable pair of glasses
* Refractive error between +8.00 D and -12.00 D, with less than 1.50 D of astigmatism

Exclusion Criteria:

* Smoker
* Pregnant or nursing
* Systemic disease that would effect tear proteins
* Punctal plugs
* Use of eye drops in the last week

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Tear protein levels | After 4-6 hours of daily wear and after one night extended wear

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Richdale, OD, PhD, Principal Investigator — State University of New York College of Optometry
Locations (1):
- SUNY College of Optometry, Clinical Vision Research Center, New York, New York, United States